CLINICAL TRIAL: NCT06626659
Title: Lipoprotein (a) and Vascular Regenerative Cell Content
Acronym: Lp(a)-VRCE
Status: Completed | Type: Observational
Sponsor: Canadian Medical and Surgical Knowledge Translation Research Group (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00080565
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Cardiovascular Diseases; Atherosclerosis Cardiovascular Disease; Ischemic Heart Disease; Dyslipidemia
Keywords: Lipoprotein (a); Progenitor cells; Cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Ischemia; Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Elevated Lp(a): Individuals with an Lp(a) level greater than or equal to 100 nmol/L
- Non-elevated Lp(a): Individuals with an Lp(a) level less than 100 nmol/L

SUMMARY:
Lp(a)-VRCE is an observational, cross sectional study looking at vessel reparative stem cell content in people with and without elevated lipoprotein (a) [Lp(a)]. Specifically, the type and number of these cells in peripheral blood samples will be measured in participants with Lp(a) ≥100 nmol/L and compared to participants with Lp(a) < 100 nmol/L. Determining the presence or absence of specific cells with blood vessel repair capacity in participants with high Lp(a) will further our knowledge of potential mechanisms through which Lp(a) influences cardiovascular health.

DETAILED DESCRIPTION:
Lipoprotein (a) [Lp(a)] is an independent, genetically determined, causal risk factor for the development of atherosclerotic cardiovascular disease. It is estimated that 20-30% of the global population have elevated Lp(a) and recent multinational guideline endorsements strongly advise the routine measuring of Lp(a), at least once in a person's life. Current Lp(a) risk level thresholds are described as <75 nmol/L for low risk and >125 nmol/L for high risk individuals. Despite ongoing clinical trials, there exists no approved therapeutic medication to specifically lower Lp(a).

Vascular regenerative cell exhaustion (VRCE) is described as the depletion of circulating pro-vascular reparative cells responsible for angiogenesis, vasculogenesis and arteriogenesis. Evidence in recent years has implicated VRCE as a novel mechanistic factor contributing to the aberrant cardiometabolic state present in type 2 diabetes, obesity, and in people of South Asian descent. It has been demonstrated that the VRCE phenotype can be reversed by treatment with sodium glucose co-transporter 2 inhibitors or bariatric surgery.

Lp(a)-VRCE is a cross-sectional, observational, two arm study enrolling 20 patients with elevated Lp(a) (≥100 nmol/L) and 20 patients with non-elevated Lp(a) (<100 nmol/L). From peripheral blood, mononuclear cells are isolated and enumerated via a multi-parametric flow cytometry assay utilizing aldehyde dehydrogenase activity and side scatter properties. The hypothesis is that people with elevated Lp(a) have comparatively different progenitor cell phenotypes to people with normal Lp(a) levels.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years of age and ≤80 years of age who meet either of the following criteria:

   1. Elevated Lp(a) (defined as greater than or equal to 100 nmol/L)
   2. Non-elevated Lp(a) (defined as less than 100 nmol/L)
2. Willing and able to provide written informed consent and comply with study procedures.

Exclusion Criteria:

1. Unable or unwilling to provide written informed consent or provide a peripheral blood sample.
2. Any life-threatening disease expected to result in death within two years of consent.
3. Any malignancy not considered cured (except basal cell carcinoma of the skin). An individual is considered cured if there has been no evidence of cancer recurrence for the five years prior to screening.
4. Uncontrolled hypertension.
5. New York Heart Association Class IV heart failure.
6. Active liver disease or liver dysfunction.
7. Active kidney disease or kidney dysfunction.
8. History of hemorrhagic stroke or other major bleeding disorder.
9. White blood cell count ≥15 x 10^9/L.
10. Women who are pregnant or nursing.
11. Previously received ribonucleic acid therapy specifically targeting Lp(a).
12. Active infectious disease requiring systemic antibiotic or anti-viral agents.
13. Known acquired immunodeficiency syndrome, such as human immunodeficiency virus.
14. On oral steroid therapy (e.g., prednisone or other corticosteroids) or other immunosuppressive agents (e.g., methotrexate).
15. Treated autoimmune disorders.
16. Participating in another study/trial that is likely to affect the primary outcome.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be identified from primary care and cardiology outpatient clinics in the Greater Toronto Area using paper-based and electronic medical records.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-10-05 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Difference in the frequency or absolute number of circulating ALDHhiSSClo primitive myeloid progenitor cells between individuals with elevated Lp(a) and individuals with non-elevated Lp(a) | Baseline

SECONDARY OUTCOMES:
Difference in the frequency/absolute count of ALDHhiSSCmid monocytes between individuals with elevated Lp(a) and individuals with non-elevated Lp(a) | Baseline

OTHER OUTCOMES:
Difference in the amount of intracellular reactive oxygen species (ROS) production in ALDHhi progenitor cell subsets | Baseline
Difference in the levels of inflammatory and oxidative stress biomarkers | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Subodh Verma, MD, Principal Investigator — University of Toronto; David A Hess, PhD, Principal Investigator — Western University, Canada
Locations (2):
- Canada (2):
  - North York Diagnostic and Cardiac Centre, North York, Ontario
  - Diagnostic Assessment Centre, Scarborough Village, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Reyes-Soffer G, Ginsberg HN, Berglund L, Duell PB, Heffron SP, Kamstrup PR, Lloyd-Jones DM, Marcovina SM, Yeang C, Koschinsky ML; American Heart Association Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Cardiovascular Radiology and Intervention; and Council on Peripheral Vascular Disease. Lipoprotein(a): A Genetically Determined, Causal, and Prevalent Risk Factor for Atherosclerotic Cardiovascular Disease: A Scientific Statement From the American Heart Association. Arterioscler Thromb Vasc Biol. 2022 Jan;42(1):e48-e60. doi: 10.1161/ATV.0000000000000147. Epub 2021 Oct 14. PMID 34647487
- [Background] Terenzi DC, Al-Omran M, Quan A, Teoh H, Verma S, Hess DA. Circulating Pro-Vascular Progenitor Cell Depletion During Type 2 Diabetes: Translational Insights Into the Prevention of Ischemic Complications in Diabetes. JACC Basic Transl Sci. 2018 Nov 5;4(1):98-112. doi: 10.1016/j.jacbts.2018.10.005. eCollection 2019 Feb. PMID 30847424
- [Background] Bakbak E, Verma S, Krishnaraj A, Quan A, Wang CH, Pan Y, Puar P, Mason T, Verma R, Terenzi DC, Rotstein OD, Yan AT, Connelly KA, Teoh H, Mazer CD, Hess DA. Empagliflozin improves circulating vascular regenerative cell content in people without diabetes with risk factors for adverse cardiac remodeling. Am J Physiol Heart Circ Physiol. 2023 Nov 1;325(5):H1210-H1222. doi: 10.1152/ajpheart.00141.2023. Epub 2023 Sep 29. PMID 37773589
- [Background] Park B, Krishnaraj A, Teoh H, Bakbak E, Dennis F, Quan A, Hess DA, Verma S. GLP-1RA therapy increases circulating vascular regenerative cell content in people living with type 2 diabetes. Am J Physiol Heart Circ Physiol. 2024 Aug 1;327(2):H370-H376. doi: 10.1152/ajpheart.00257.2024. Epub 2024 Jun 14. PMID 38874618
- [Background] Krishnaraj A, Bakbak E, Teoh H, Pan Y, Firoz IN, Pandey AK, Terenzi DC, Verma R, Bari B, Bakbak AI, Kunjummar SP, Yanagawa B, Connelly KA, Mazer CD, Rotstein OD, Quan A, Bhatt DL, McGuire DK, Hess DA, Verma S. Vascular Regenerative Cell Deficiencies in South Asian Adults. J Am Coll Cardiol. 2024 Feb 20;83(7):755-769. doi: 10.1016/j.jacc.2023.12.012. PMID 38355246
- [Background] Kronenberg F, Mora S, Stroes ESG, Ference BA, Arsenault BJ, Berglund L, Dweck MR, Koschinsky M, Lambert G, Mach F, McNeal CJ, Moriarty PM, Natarajan P, Nordestgaard BG, Parhofer KG, Virani SS, von Eckardstein A, Watts GF, Stock JK, Ray KK, Tokgozoglu LS, Catapano AL. Lipoprotein(a) in atherosclerotic cardiovascular disease and aortic stenosis: a European Atherosclerosis Society consensus statement. Eur Heart J. 2022 Oct 14;43(39):3925-3946. doi: 10.1093/eurheartj/ehac361. PMID 36036785
- [Derived] Moroney M, Casey JH, Teoh H, Krishnaraj A, Pan Y, Quan A, Patel SK, Dennis F, He AZ, Park B, Verma R, Misner E, Seguchi R, Hassan SMA, Dennis CJ, Meglis G, Pandey A, Butler J, Mazer CD, Byrne RA, Koschinsky ML, Hess DA, Verma S. Vascular regenerative deficiencies in people with elevated lipoprotein(a): the Lp(a)-VRCE CardioLink-16 translational study. Cardiovasc Res. 2025 Nov 22;121(14):2127-2130. doi: 10.1093/cvr/cvaf142. PMID 40883226